CLINICAL TRIAL: NCT06896240
Title: The Impact of a Daily Whole Food Plant-based Smoothie Utilization 2 Weeks Prior to Revision Total Knee Replacement Surgery on Inflammation and Post-operative Pain.
Brief Title: Fiber Smoothie Supplement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-2396
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Total Knee Arthroplasty Revision; Inflammatory Markers; Gut Microbiota
Keywords: TKA Revision; Inflammation; Diet; Gut Microbiome
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: A randomized control trial of two groups, intervention vs. control.
Who Masked: Outcomes Assessor
Masking Description: Primary investigator will be blinded from which group participants are blinded from. Participants will be aware of what group they are in because they will be required to take the smoothie intervention before surgery. The RA will perform randomization and has to complete smoothie compliance calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 No Smoothie (No Intervention): This group will make no changes to their pre-operative diet and will not consume the smoothie leading up to their TKA revision surgery.
- Group 2 Smoothie (Experimental): This group will receive the "Green Smoothie Guide" from the American College of Lifestyle Medicine which they will use to prepare a daily smoothie for the 14 days leading up to their total knee arthroplasty revision surgery. No other changes will be made to their pre-operative diet.
  Interventions: Dietary Supplement: Assigned Interventions

INTERVENTIONS:
Dietary Supplement: Assigned Interventions — The "Green Smoothie Guide" from the American College of Lifestyle Medicine contains guidelines for a 6-step smoothie to include whole and high fiber foods.
  Arms: Group 2 Smoothie

SUMMARY:
This study aims to assess the feasibility of a 2-week dietary whole-food smoothie intervention and compare outcomes between two groups: patients that integrated a daily whole food plant-based smoothie into their diet for two weeks prior to surgery, and a control group of revision TKA patients that made no nutritional changes to their diet prior to surgery. The main research questions are:

1. Among patients planned for elective TKA revision surgery, what is the feasibility of a 2-week dietary intervention implemented 2 weeks prior to surgery? [Outcomes will be compliance, noted barriers and/or facilitators, satisfaction with diet]
2. Determine if the implementation of a daily whole food plant- based smoothie dietary supplement 2 weeks prior to TKA revision surgery will reduce inflammation -measured in plasma levels of IL-6 and CRP- at POD0, POD1, POD2, POD3, and 6 Weeks Post-operative as compared to 1) baseline (prior to dietary intervention initiation) and 2) control patients who did not make changes in their diet prior to surgery.
3. Determine if the implementation of a daily whole food plant-based smoothie dietary supplement 2 weeks prior to TKA revision surgery will result in quantifiable changes in the gut microbiome composition -measured via fecal samples- as compared to control patients who did not make changes in their diet prior to surgery.
4. Determine if the implementation of a daily whole food plant- based smoothie dietary supplement 2 weeks prior to TKA revision surgery will result in improved immediate postoperative pain -measured through numeric rating scale (NRS) pain scores- and opioid use -measured in morphine milligram equivalents (MME)- as compared to control patients.
5. Compare patient satisfaction and adoption of nutritional behavioral changes in patients implementing a whole food plant-based smoothie 2 weeks prior to TKA revision surgery to patients undergoing the same surgery but did not me pre-surgery dietary changes.

The researcher's primary outcome is measuring feasibility and patient compliance with smoothie consumption. Secondarily, the investigators are interested in measuring if the preoperative smoothie can alter the gut microbiome and decrease systemic inflammation, leading to lowered post-operative pain and opioid use.

DETAILED DESCRIPTION:
This study aims to assess the feasibility of a 2-week dietary whole-food smoothie intervention and compare outcomes between two groups: patients that integrated a daily whole food plant-based smoothie into their diet for two weeks prior to surgery, and a control group of revision TKA patients that made no nutritional changes to their diet prior to surgery. The main research questions are:

1. Among patients planned for elective TKA revision surgery, what is the feasibility of a 2-week dietary intervention implemented 2 weeks prior to surgery? [Outcomes will be compliance, noted barriers and/or facilitators, satisfaction with diet]
2. Determine if the implementation of a daily whole food plant- based smoothie dietary supplement 2 weeks prior to TKA revision surgery will reduce inflammation -measured in plasma levels of IL-6 and CRP- at POD0, POD1, POD2, POD3, and 6 Weeks Post-operative as compared to 1) baseline (prior to dietary intervention initiation) and 2) control patients who did not make changes in their diet prior to surgery.
3. Determine if the implementation of a daily whole food plant-based smoothie dietary supplement 2 weeks prior to TKA revision surgery will result in quantifiable changes in the gut microbiome composition -measured via fecal samples- as compared to control patients who did not make changes in their diet prior to surgery.
4. Determine if the implementation of a daily whole food plant- based smoothie dietary supplement 2 weeks prior to TKA revision surgery will result in improved immediate postoperative pain -measured through numeric rating scale (NRS) pain scores- and opioid use -measured in morphine milligram equivalents (MME)- as compared to control patients.
5. Compare patient satisfaction and adoption of nutritional behavioral changes in patients implementing a whole food plant-based smoothie 2 weeks prior to TKA revision surgery to patients undergoing the same surgery but did not me pre-surgery dietary changes.

Participants will be randomly assigned to consume the whole food plant-based smoothie intervention daily for the two weeks leading up to surgery, or to have no preoperative diet intervention (control group).

The researcher's primary outcome is measuring feasibility and patient compliance with smoothie consumption. Secondarily, the investigators are interested in measuring if the preoperative smoothie can alter the gut microbiome and decrease systemic inflammation, leading to lowered post-operative pain and opioid use.

ELIGIBILITY:
Inclusion:

* Scheduled for revision TKA at HSS with participating surgeons; not as a result of infection or trauma and all components (tibial and femoral) needing replacement
* Age between 40 and 80
* Diagnosed with osteoarthritis
* Diagnosed with 2+ modifiable chronic lifestyle diseases: Type 2 DM, CVD (such as CAD, heart disease, stroke, HTN), stress, anxiety, depression, ADHD, metabolic syndrome, certain types of cancer (such as breast, colorectal, lung, prostate), Alzheimer's disease, vascular cognitive impairment, CKD, RA, asthma, chronic pain conditions (such as chronic back pain and osteoarthritis), fibromyalgia, migraines, COPD (Steiber 2011, Grant 2014)
* ASA Class 1 ('normal' healthy patient) or 2 (patient with mild systemic disease and no functional limitations; the diseases the patient has are well controlled)
* Ability to understand written and spoken English
* Willing to complete entire pre-operative and post-operative work up in NYC, main campus site
* Willing to follow a 2-week smoothie supplement, including willingness to purchase ingredients and have access to a blender for preparation

Exclusion:

* Age >80 years or <40 years
* Revision due to infection or trauma
* ASA class 3 (patient with severe systemic disease that results in functional limitations) or 4 (patient with severe systemic disease that is a constant threat to life)
* Not interested or unable to provide informed consent
* Unstable weight (>5kg weight change in the past 3 months, documented in Epic) or currently on weight loss drugs such as GLP-1 agonists (Prasad et al., Cardiovasc Diabetol 2022; empagliflozin CRP studies.)
* Active infection, flare-up of seasonal allergies, or physical trauma (all can alter CRP)
* Medication changes the month leading up to surgery
* Specifically medications altering inflammation: Statins (Ridker 2008), steroids (Boumpas et al., Ann Intern Med 1993; glucocorticoid cytokine modulation research.), DMARDS/biologics/immunosuppressants (Clinical rheumatology guidelines, biologic RCTs (e.g., TNF inhibitors, IL-6 inhibitors), Colchicine (Tardif et al., N Engl J Med 2019; colchicine cardiovascular inflammation studies.), hormone replacement therapies (Ridker et al., JAMA 1999; OCs and CRP meta-analyses.), new psychiatric medications (Miller & Raison, Nat Rev Immunol 2016; psychotropic-inflammation associations.)
* BMI >40 kg/m2
* Food intolerance/allergy/sensitivity to ingredients suggested for smoothies
* History of IBD (and IBD medication)
* History of bariatric surgery
* History of cancer
* History of thyroid disease
* History of or current drug abuse
* Pregnancy
* Current smoker
* Any patient with an electronic cardiac implant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Measured in Terms of Compliance | Daily for 14 days pre-operative
  Compliance is measured as number of days in the two-week intervention timeframe that patients reported having consumed the smoothie. The investigators will conduct fourteen daily phone calls to assess yes/no smoothie intake and ingredients used. Informed by nutrition compliance in the literature, the investigators will apply an 80% threshold for compliance rate which translates to roughly 11/14 days. The compliance range is 0%-100% or 0-14 days with 100% or 14 days indicating higher smoothie compliance and a more favorable outcome.
Feasibility Measured in Terms of Noted Barriers/Facilitators | Day 0
  Noted barriers/facilitators are open-ended questions in unstructured free text format. A feedback form will be sent to participants, and feedback and suggestions will be recorded by the investigators.
Feasibility Measured in Terms of Satisfaction with Diet | Baseline and 6 weeks post-operative
  The quantification of satisfaction with diet using the verified Diet Satisfaction Scale with 28 questions. Individual questions are scored on a scale of 1-5 with a higher score indicating higher diet satisfaction and a more favorable outcome. Scores from each question will be compiled into a total score for the questionnaire.

SECONDARY OUTCOMES:
Inflammation and Pain Control: C-Reactive Protein | Baseline, Day 0, Day 1, Day 2, Day 3, 6 weeks post-op
  Inflammation and pain control are quantified by biological markers of inflammation such as C-reactive protein found in the blood. C-reactive protein is produced in the liver, and its levels rise in response to inflammation. A normal range of C-reactive protein is less than 0.3mg/dL and is a more favorable outcome than an elevated level of C-reactive protein.
Inflammation and Pain Control: Interleukin 6 | Baseline, Day 0, Day 1, Day 2, Day 3, 6 weeks post-op
  Inflammation and pain control are quantified by biological markers of inflammation such as the pro-inflammatory cytokine, interleukin 6, found in the blood. An elevated amount of Interleukin 6, above 15pg/mL, is indicative of increased inflammatory response in the body and is less favorable outcome.
Inflammation and Pain Control: Microbiome Composition | Baseline, 4 Days Pre-op, 2 Days Pre-op
  Inflammation and pain control are quantified firstly by biological markers of inflammation such as microbiome composition. Participants will complete three self-administered stool sample collections and ship their samples to Mount Sinai Laboratory. Mount Sinai will conduct raw 16S rRNA sequencing to show alpha and beta bacteria diversity. Higher diversity 4 days pre-op and 2 days pre-op relative to baseline is indicative of a more successful intervention and a more favorable outcome.
Inflammation and Pain Control- Numerical Rating Scales | Baseline, Day 0, Day 1, Day 2, Day 3, 6 weeks post-op
  Inflammation and pain control are quantified firstly by markers of acute pain/analgesia which are measured by Numerical Rating Scales (NRS) of pain. Participants will be asked questions about their knee pain on a scale of 0-10 where higher scores are indicative of increased pain and a less favorable outcome.
Inflammation and Pain Control: Opioid Intake | Postoperatively; 0-24 hours, 24-48 hours, and 48-72 hours
  Inflammation and pain control are quantified by markers of acute pain/analgesia such as opioid intake. Opioid intake will be recorded from participants' medical charts while they are under care at HSS Main Hospital. Opioid intake will be measured in morphine milligram equivalents (MME) with a lower opioid intake being more favorable.
Diet Quantification | Baseline, Day 0, and 6 weeks post-op.
  Diet will be quantified using Diet ID Inc.'s online software, a validated tool, which measures diet quality, caloric intake, and nutrient intake. After participants go through the Diet ID survey, the Diet ID platform will calculate a "Nutrition Score" which will be the recorded value of nutrition. The scores will be reported on a scale of 1-10 with higher scores indicating "better" nutrition and a more favorable outcome.
BIA Measurements: Phase Angle | Baseline, Day 0, and 6 weeks post-op.
  Bioelectrical Impedance Analysis (BIA) produces a measurement of phase angle (PhA) which measures the water distribution among intracellular and extracellular space. Phase angle is measured in degrees with 6.5-7.5 degrees being described as a healthy range and lower degrees being less favorable.
BIA Measurements: Fat-Free Mass (Index) | Baseline, Day 0, and 6 weeks post-op.
  Bioelectrical Impedance Analysis (BIA) produces a measurement of fat-free mass (FFM) which is a measurement of the total body weight excluding fat. BIA testing produces a fat-free mass weight in kg which is divided by the total kg of the participant to produce a percentage of fat-free mass. For men, a healthy range for a fat-free mass percentage is ~78%-87%, and for women, a healthy range is ~67%-75%. The fat-free mass index measurement can also be calculated using the measurement of fat-free mass relative to height.
BIA Measurements: Extracellular Water | Baseline, Day 0, and 6 weeks post-op.
  Bioelectrical Impedance Analysis (BIA) can produce measurements of extracellular water (ECW) which is the water outside of the cells.
BIA Measurements: Extracellular Water, Total Body Water, and Ratio ECW/TBW | Baseline, Day 0, and 6 weeks post-op.
  Bioelectrical Impedance Analysis (BIA) can produce measurements of Extracellular Water (ECW)--the fluid outside of the cells--and Total Body Water (TBW). Then, a ratio of extracellular water to total body water (ECW/TBW) can be calculated with a normal range for this ratio being 0.360-0.390. A higher value for this ratio is indicative of a less favorable outcome.
PROMIS-Global 10 | Baseline, Day 0, 6 weeks post-op, and 6 months post-op.
  The PROMIS-Global 10 is a validated 10-item questionnaire to evaluate health in relation to quality of life. Questions are rated on a scale of 1-5 with a higher score being indicative of higher health and a more favorable outcome. Scores for all questions will be added up to calculate a total score.
Range of Motion | Baseline, Day 0, Day 1, Day 2, Day 3, 6 weeks post-op
  Angle of knee movement in degrees as recorded during all standard of care visits. Measurement points include: the internist physician during pre-surgical screening, the surgeon on Day 0, physical therapy on Days 1-3, the surgeon during the 6-week post-operative follow-up visit.
Frailty | Baseline
  The 5-Item frailty index is a standardized, comorbidity-based risk stratification tool used to predict adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Tafuro, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- HSS Main Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No